CLINICAL TRIAL: NCT04331600
Title: Multicenter, Randomized, Open-label, Non-commercial, Investigator-initiated Study to Evaluate the Efficacy and Safety of Chloroquine Phosphate in Combination With Telemedicine Care in the Risk Reduction of COVID-19 Related Hospitalization or Death, in Ambulatory Patients With COVID-19 Being at Risk of Serious Complications
Brief Title: Chloroquine as Antiviral Treatment in Coronavirus Infection 2020
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WROCLAW CORONA STUDY 2020
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — chloroquine diphosphate; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHLOROQUINE (Experimental): Standard of care + chloroquine phosphate + telemedical approach.
  Interventions: Drug: Chloroquine phosphate; Other: Telemedicine
- CONTROL GROUP (Other): Standard of care + telemedical approach.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Drug: Chloroquine phosphate — Oral chloroquine phosphate for 14 days
  Arms: CHLOROQUINE
Other: Telemedicine — Telemedical supervision for 42 days

SUMMARY:
The aim of the study is to evaluate whether the therapy with chloroquine phosphate (CQ, in combination with telemedical approach) in addition to standard care is effective and safe in reducing composite endpoint of COVID-19-related hospitalization or all cause death, in ambulatory patients with SARS-SoV-2 infection at particular risk of serious complications due to advanced age and/or comorbid conditions (in comparison with subjects not treated with CQ but receiving standard care and supervised telemedically).

DETAILED DESCRIPTION:
Until now there are no evidence-based, good-quality data from sufficiently powered clinical trials supporting the use of any antiviral medicines or immunomodulatory therapies in the management or prophylaxis of COVID-19; however there are currently being initiated studies in Europe and U.S., and a few registered studies are ongoing in China. Currently two groups of medicines are hypothesized to be effective therapeutic options in COVID-19: (1) classical antiviral drugs interfering with pathogen dissemination / replication, and (2) compounds inhibiting host inflammatory reactions, especially (and potentially selectively) in respiratory tract / system (cytokine inhibitors and specific antibodies). Special hopes are placed in quinoline derivatives such as chloroquine (CQ), based on some unpublished data from China and a few experiments in vitro. CQ is an old antimalarial drug that has been used for more than 50 years in the therapy and prevention of this parasitosis. Anti-inflammatory features of quinolone derivatives such as CQ or hydroxychloroquine have also been used in rheumatology (for the therapy of lupus erythematosus or rheumatoid arthritis) due to the inhibition of the production of proinflammatory cytokines. The effectiveness (and safety) of CQ in COVID-19 has not been investigated in sufficiently powered RCTs until now.

ELIGIBILITY:
INCLUSION CRITERIA

1. age >=60 years OR age 18-59 years with one of the following conditions:

   1. chronic lung disease
   2. chronic cardiovascular disease
   3. diabetes
   4. malignancy diagnosed within 5 years prior to enrollment
   5. history of chronic kidney disease
   6. atrial fibrillation
   7. past haemorrhagic stroke, ischemic stroke or transient CNS ischemia
   8. obesity defined as BMI ≥ 30 kg / m2
   9. 10-year risk of fatal cardiovascular disease
2. SARS-CoV-2 infection confirmed in RT-PCR (nasopharyngeal swab)
3. Hospitalization not required based on clinical judgement
4. Ability to participate in telemedical care

EXCLUSION CRITERIA

1. Lack of written informed consent
2. Possible failure to comply with the protocol
3. Chloroquine, hydroxychloroquine therapy within 30 days prior to enrollment
4. Antiviral therapy within 14 days prior to enrollment
5. Contraindications to chloroquine (pregnancy, breast-feeding, severe renal insufficiency, amiodarone therapy, alcohol disease, haematological disorders, epilepsia, porphyria, liver disease/cirrhosis, retinopathy, fainting/syncope, myasthenia)
6. Hypersensitivity to chloroquine or drug excipients
7. HIV infection
8. Other relevant circumstances/conditions based on clinical judgement
9. Concurrent participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
COVID-19-related hospitalization or all-cause death | 15 days
  Composite endpoint of COVID-19-related hospitalization or all-cause death

SECONDARY OUTCOMES:
Decrease in COVID-19 symptoms | 15 days and 42 days
  Decrease in self-reported symptoms of novel coronavirus infection. Non-dichotomous symptoms (e.g. syncope is dichotomous - yes or no) such as dyspnoea will be self-evaluated by patients using the 0-3 scale with the severity increasing with the punctation (0-no symptoms, 1-mild symptoms, 2-moderate symptoms, 3-severe symptoms).
Development of pneumonia | 42 days
  Based on X-ray, microbiology and laboratory results
Development of coronavirus infection-related complications | 42 days
  Acute respiratory distress syndrome, bacterial infection, shock, sepsis, etc

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Uniwersytecki Szpital Kliniczny, Wroclaw, Ul. Borowska 213
  - Wielospecjalistyczny Szpital Miejski, Poznan, Ul. Szwajcarska 3

IPD SHARING:
Plan to Share IPD: No